CLINICAL TRIAL: NCT01648543
Title: Comparison of Methods of Lumbar Sympathetic Ganglion Block: Distance vs Angle
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, jong bum Choi, Yonsei University College of Medicine, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3-2012-0042
Record Dates: First submitted 2012-07-19; First posted 2012-07-24 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-07

CONDITIONS: Lumbar Sympathetic Ganglion Block Indication: Neuropathic Pain, CRPS, Hyperhydrosis Etc.

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- block method: angle (Active Comparator): The entry angle of angular method which is one method of lumbar sympathetic ganglion block is 30 degree of anterior-posterior view of C-arm.
  Interventions: Procedure: lumbar sympathetic ganglion block
- block method: distance (Active Comparator): The entry point of modified Reid method which is popular method of lumbar sympathetic ganglion block is 7~7.5cm from midline of spinous process of lumbar spine.
  Interventions: Procedure: lumbar sympathetic ganglion block

INTERVENTIONS:
Procedure: lumbar sympathetic ganglion block

SUMMARY:
Lumbar sympathetic ganglion block is used for several neuropathic pain syndromes. The best method of lumbar sympathetic ganglion block is not established. The investigators would compare two methods of lumbar sympathetic ganglion block. One is modified Reid method which's entry point is 7~7.5cm from midline of spinous process of lumbar spine. The other is angular method which's entry angle is 30 degree from anterior-posterior view of C-arm. Comparison modified Reid method with angular method would be helpful for finding best method of lumbar sympathetic ganglion block.

ELIGIBILITY:
Inclusion Criteria:

1. Adults above age of 20
2. Undergoing lumbar sympathetic ganglion block indication

Exclusion Criteria:

1. Infection
2. Bleeding tendency
3. Previous spinal surgery history
4. Pregnancy
5. Illiteracy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2012-06; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
temperature change | 30min
muscle or vessel shadow | 30min

CONTACTS AND LOCATIONS:
Overall Officials: Jong Bum Choi, Study Director — Yonsei University
Locations (1):
- Gangnam Severance Hospital, Seoul, South Korea